CLINICAL TRIAL: NCT04547153
Title: Infusional Fluorouracil and Weekly Docetaxel as First-line Therapy for Gastric Cancer With Bone Marrow Metastasis and Disseminated Intravascular Coagulation: a Multi-center, Phase II Trail
Brief Title: Infusional Fluorouracil and Weekly Docetaxel for Gastric Cancer With Bone Marrow Involvement and DIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, MD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhenLong
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer; Bone Marrow Metastasis; Disseminated Intravascular Coagulation
Keywords: 5-fluorouracil; docetaxel
MeSH Terms: conditions — Stomach Neoplasms; Disseminated Intravascular Coagulation | interventions — Fluorouracil; Docetaxel; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LD-FUD (Zhen Long) (Experimental): 5-fluorouracil 200mg/square metre/day continuously venous infusion on days 1-21; Docetaxel 25mg/square metre, on days 1, 8 and 15; This regimen repeats every 4 weeks.
  Interventions: Drug: 5-fluorouracil; Drug: Docetaxel

INTERVENTIONS:
Drug: 5-fluorouracil — 200mg/square metre/day civ D1-D21
  Other Names: 5-Fu
Drug: Docetaxel — 25mg/square metre ivdrip D1, D8, D15
  Other Names: D

SUMMARY:
A distinctive subtype of gastric adenocarcinoma with extensive bone marrow metastasis and DIC has been described. Few patients have been treated properly due to the lack of standard care. We designed this phase II study to evaluate a dose-dense regimen for this kind of highly aggressive gastric cancer (HAGC).

DETAILED DESCRIPTION:
5-fluorouracil 200mg/square metre/day continuously venous infusion on days 1-21; Docetaxel 25mg/square metre, on days 1, 8 and 15; This regimen repeats every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-3;
* Pathologically confirmed adenocarcinoma in stomach or esophagogastric junction;
* Bone marrow metastasis confirmed by aspiration, biopsy or PET/CT scan;
* overt DIC according to the International Society on Thrombosis and Haemostasis (ISTH) criteria;
* Treatment-naive after the diagnosis of metastasis;
* Platelet ≤ 50 * 10E9/L;
* ALT≤5×ULN, AST≤5×ULN, Bilirubin≤5×ULN, Creatinine≤3×ULN;
* Written informed consent.

Exclusion Criteria:

* Concurrent aggressive malignancy;
* Docetaxel containing perioperative treatment within 6 months;
* Allergic to the study drugs;
* Serious medical conditions, including severe heart disease, severe cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection,etc.
* HIV positive;
* MSI-H;
* Her-2 gene overexpression;
* Inadequate contraceptive measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
hematological response rate (HeRR) | 2 months
  percentage of participants whose platelet restored to normal range

SECONDARY OUTCOMES:
time to hematological response (TTHeR) | 2 months
  the interval from treatment to hematological response
one-month mortality (OMM) | 30 days
  the proportion of participants who die within 30 days after the chemotherapy
overall survival (OS) | 2 years
  from the start of chemotherapy to the date of death of any cause or censored at the last date known to be alive
toxicities | 2 months
  in terms of incidence of adverse events, according to the National Cancer Institute Common Toxicity Criteria version 5.0
quality of life assessed by EORTC QOL C-30 and STO-22 (QoL) | 3 months
  individual QoL based on questionnaire scores change from baseline to experimental treatment end and 28-day post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Jian Xiao, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: July 2024 - June 2027
Access Criteria: Researchers interested in the same disease

REFERENCES:
- [Background] Morita R, Ishikawa T, Sawai Y, Kajiwara M, Asaeda K, Kobayashi R, Miyazaki H, Doi T, Inoue K, Dohi O, Yoshida N, Kamada K, Uchiyama K, Takagi T, Konishi H, Naito Y, Itoh Y. [A Long-Term Survival Case of Gastric Cancer with Disseminated Intravascular Coagulation due to Myelocarcinomatosis Treated with S-1 plus Oxaliplatin Therapy]. Gan To Kagaku Ryoho. 2021 May;48(5):731-734. Japanese. PMID 34006725
- [Background] Kwon JY, Yun J, Kim HJ, Kim KH, Kim SH, Lee SC, Kim HJ, Bae SB, Kim CK, Lee NS, Lee KT, Park SK, Won JH, Hong DS, Park HS. Clinical outcome of gastric cancer patients with bone marrow metastases. Cancer Res Treat. 2011 Dec;43(4):244-9. doi: 10.4143/crt.2011.43.4.244. Epub 2011 Dec 27. PMID 22247710
- [Derived] Xiaohui Z, Shanshan L, Taiyuan C, Ge D, Hongen Y, Lishuo S, Xiaoru L, Wanjia H, Jian X. Docetaxel and fluorouracil as first-line therapy for gastric cancer with bone marrow metastasis and disseminated intravascular coagulation. Future Oncol. 2022 Nov;18(35):3875-3880. doi: 10.2217/fon-2022-0748. Epub 2022 Nov 8. PMID 36346044